CLINICAL TRIAL: NCT01618149
Title: Use Dual-energy X-ray Absorptiometry and Quantitative Microradiography to Predict the Periprosthetic Bone Loss in Distal Femur After Total Knee Arthroplasty
Brief Title: Use Quantitative Microradiography to Predict the Periprosthetic Bone Loss in Distal Femur After Total Knee Arthroplasty
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor-Investigator, National Taiwan University Hospital, Use dual-energy x-ray absorptiometry and quantative microradiography to predict the periprosthetic bone loss in distal femur after total knee arthroplasty, National Taiwan University Hospital
Other Study IDs: 201204035RIB
Record Dates: First submitted 2012-06-11; First posted 2012-06-13 (Estimated); Last update posted 2012-06-13 (Estimated); Status verified 2012-06

CONDITIONS: Periprosthetic Bone Loss in Total Knee Replacement
Keywords: osteoarthritis; periprosthetic bone loss; dual energy x-ray absorptiometry
MeSH Terms: conditions — Osteoarthritis | interventions — Absorptiometry, Photon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A 2X1X0.5cm bone fragment harvested during the chamfer cut of total knee arthroplasty
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- severe knee OA who are indicated for total knee arthroplasty: the woman who are indicated for TKR and are post menopausal will be recruited in this study. We will excluded the patients who had immune disease ,previous fracture of femur and end stage of renal disease
  Interventions: Radiation: dual energy x-ray absorptiometry

INTERVENTIONS:
Radiation: dual energy x-ray absorptiometry — before the surgery of total knee arthroplasty and after the surgery 6 months and 12 months

SUMMARY:
The investigators hypothesized that the microarchitecture of bone influence the degree of periprosthetic bone loss after total knee arthroplasty surgery. The investigators collected the bone fragment at the distal femur while performing total knee replacement and take quantitative radiography analysis . Before and after the surgery(6 month ,12 month) , the investigators check the BMD at identical location of the distal femur by using dual energy absorptiometry. The investigators will use linear regression to evaluate the relationship between the microarchitecture and the degree of bone loss.

ELIGIBILITY:
Inclusion Criteria:

* severe knee osteoarthritis
* post menopausal women

Exclusion Criteria:

* immune disease
* end stage of renal disease who receive dialysis
* history of fracture at ipsilateral distal femur

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the patients who are indicated for total knee arthroplasty and are post menopausal women. The patients who had history of immune disease , fracture of the femur and end stage of renal disease will be excluded
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2012-07; Primary Completion 2013-07 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
change in bone mineral density | before the surgery and after the sugery (6month ,12month)
  Use dual energy x-ray absorptiometry to detect to BMD at the distal femur

CONTACTS AND LOCATIONS:
Overall Officials: ching chuan Jiang, professor, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National taiwan university hospital, Taipei, Taiwan, Taiwan